CLINICAL TRIAL: NCT00018616
Title: Improving Compliance With Metformin
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Rosen, Marc - Principal Investigator, Department of Veterans Affairs
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: MHBS-047-98F
Record Dates: First submitted 2001-07-03; First posted 2001-07-05 (Estimated); Last update posted 2009-09-23 (Estimated); Status verified 2009-09

CONDITIONS: Diabetes
Keywords: compliance; MEMS; metformin
MeSH Terms: conditions — Diabetes Mellitus; Patient Compliance

ARMS (1):
- 1 (Other)
  Interventions: Behavioral: MEMS caps

INTERVENTIONS:
Behavioral: MEMS caps

SUMMARY:
This is a randomized controlled trial of adherence. The study involves monitoring and managing focused intervention in patients prescribed metformin.

DETAILED DESCRIPTION:
The active intervention, MEMS Feedback, involves review of patients' medication-taking over the preceding weeks

ELIGIBILITY:
Inclusion Criteria:

* Metformin has been prescribed
* Willing to use medication containers with MEMS caps
* Capable of giving informed consent

Exclusion Criteria:

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 79 (Actual)
Dates: Start 1999-10; Primary Completion 2004-01 (Actual); Study Completion 2005-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marc I. Rosen, MD, Principal Investigator — VA Connecticut Health Care System (West Haven)
Locations (1):
- VA Connecticut Health Care System (West Haven), West Haven, Connecticut, United States